CLINICAL TRIAL: NCT00941889
Title: The Effect of Human Papillomavirus Vaccination on Recurrence Rates in HIV Positive Patients Treated for Anal Condylomata
Brief Title: The Effect of HPV Vaccination on Recurrence Rates in HIV Patients With Condylomata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HRPO 07-0648
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: HIV Positive; Anal Condylomata; Anal Warts; HIV Infections
Keywords: HIV; HPV; Anal condylomata; Vaccine; HIV positive patients; Anal condylomata or anal warts
MeSH Terms: conditions — HIV Seropositivity; HIV Infections | interventions — Sodium Chloride; Vaccines, Synthetic; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Patients who are in the control group received a placebo of saline in the upper extremity at initial visit, 2 months and 6 months after enrollment.
  Interventions: Drug: Saline
- Gardasil (Active Comparator): The treatment group received a 0.5mL intramuscular injection of Gardasil (quadrivalent HPV vaccine) in their upper extremity at initial visit, and again at two months and six months after enrollment.
  Interventions: Drug: Quadrivalent Human Papillomavirus (Types 6,11,16,18) Recombinant Vaccine

INTERVENTIONS:
Drug: Saline — 0.5 ml
  Arms: Placebo
Drug: Quadrivalent Human Papillomavirus (Types 6,11,16,18) Recombinant Vaccine — 0.5mL intramuscular injection of Gardasil (quadrivalent HPV vaccine) in their upper extremity initially and again at two months and six months after enrollment.
  Other Names: GARDASIL
  Arms: Gardasil

SUMMARY:
The primary objective of this pilot study is to evaluate the effect of the HPV vaccine Gardasil on anal condylomata recurrence and persistence rates in HIV positive patients.

DETAILED DESCRIPTION:
A quadrivalent human papilloma virus (HPV) vaccine called Gardasil had recently (at start of study) been developed and approved by the FDA for the prevention of cervical HPV infection and cervical cancer, which is associated with infection from this virus. It is unknown whether the same vaccine could also be of benefit in treating anogenital warts, which are caused by the same virus. This is an important and clinically relevant question which needs to be answered. Anal warts have a high prevalence and recurrence and usually require extended lengths of treatment and follow-up, especially in the HIV population. At times, treatment of anal warts requires multiple surgeries to excise them if the burden of disease is high. Therefore, this disease represents a significant expense to patients and the health care system.

Further, the HPV virus that causes anal warts has been associated with anal cancer and with its preliminary lesion known as anal intraepithelial neoplasia (AIN). This study touches on two important, relevant and costly healthcare issues: finding a better treatment for the most common sexually transmitted disease in our country, and helping to prevent anal cancer, which is often a fatal disease.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age;
* HIV positive status;
* CD4 > 200 and viral RNA < 400 on anti-retroviral therapy (HAART) or CD4 > 350 if not on HARRT;
* the presence of anal warts that require surgical excision/ablation.

Exclusion Criteria:

* CD4 < 200 and/or viral RNA > 400 on HAART or CD4 < 350 and not on HAART ;
* low burden of anal warts that would not require surgical excision/ablation;
* previous vaccinations against HPV or allergic reactions to any vaccine component;
* patients who are currently pregnant;
* patients with a previous diagnosis of anal cancer;
* patients who are incarcerated;
* patients who have taken immunomodulators (i.e. interferon, interleukin, corticosteroids, etc.) within the last 90 days;
* patients who have had an opportunistic infection in the last 90 days or who have another intercurrent illness that precludes their safe enrollment in this study;
* patients who, in the judgment of the investigators, are unlikely to adhere to the protocol, either because of a substance abuse or psychiatric diagnosis, or other factors that would affect compliance;
* failure to strictly comply with the vaccination schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Hunt, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, Section of Colon Rectal Surgery, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
No outcomes data were collected or analyzed due to lack of participant follow-up.

REFERENCES:
- [Background] StatBite: Prevalence of HPV in a cohort of U.S. men. J Natl Cancer Inst. 2009 Feb 18;101(4):223. doi: 10.1093/jnci/djp008. Epub 2009 Feb 10. No abstract available. PMID 19211451
- [Background] Human papillomavirus vaccines. WHO position paper. Wkly Epidemiol Rec. 2009 Apr 10;84(15):118-31. No abstract available. English, French. PMID 19360985
- [Background] Chitale R. Merck hopes to extend gardasil vaccine to men. J Natl Cancer Inst. 2009 Feb 18;101(4):222-3. doi: 10.1093/jnci/djp014. Epub 2009 Feb 10. No abstract available. PMID 19211446
- [Background] Gillespie MB, Smith J, Gibbs K, McRackan T, Rubinchik S, Day TA, Sutkowski N. Human papillomavirus and head and neck cancer: a growing concern. J S C Med Assoc. 2008 Dec;104(8):247-51. PMID 19326612
- [Background] Stanley M. The epidemiology and burden of HPV disease. Nurs Times. 2008 Sep 9-15;104(36):38-40. PMID 18822547
- [Background] Gross G. Impact of prophylactic human papillomavirus vaccines on dermatology and venereology. G Ital Dermatol Venereol. 2008 Aug;143(4):259-65. PMID 18833082
- [Background] Herbert J, Coffin J. Reducing patient risk for human papillomavirus infection and cervical cancer. J Am Osteopath Assoc. 2008 Feb;108(2):65-70. PMID 18303060
- [Background] Dowling TS. Mandating a human papillomavirus vaccine: an investigation into whether such legislation is constitutional and prudent. Am J Law Med. 2008;34(1):65-84. doi: 10.1177/009885880803400103. No abstract available. PMID 18512537
- [Background] Dunne EF, Markowitz LE. Genital human papillomavirus infection. Clin Infect Dis. 2006 Sep 1;43(5):624-9. doi: 10.1086/505982. Epub 2006 Jul 26. PMID 16886157
- [Background] Winer RL, Lee SK, Hughes JP, Adam DE, Kiviat NB, Koutsky LA. Genital human papillomavirus infection: incidence and risk factors in a cohort of female university students. Am J Epidemiol. 2003 Feb 1;157(3):218-26. doi: 10.1093/aje/kwf180. PMID 12543621
- [Background] Vukasin P. Anal condyloma and HIV-associated anal disease. Surg Clin North Am. 2002 Dec;82(6):1199-211, vi. doi: 10.1016/s0039-6109(02)00085-3. PMID 12516848
- [Background] Villa LL, Costa RL, Petta CA, Andrade RP, Ault KA, Giuliano AR, Wheeler CM, Koutsky LA, Malm C, Lehtinen M, Skjeldestad FE, Olsson SE, Steinwall M, Brown DR, Kurman RJ, Ronnett BM, Stoler MH, Ferenczy A, Harper DM, Tamms GM, Yu J, Lupinacci L, Railkar R, Taddeo FJ, Jansen KU, Esser MT, Sings HL, Saah AJ, Barr E. Prophylactic quadrivalent human papillomavirus (types 6, 11, 16, and 18) L1 virus-like particle vaccine in young women: a randomised double-blind placebo-controlled multicentre phase II efficacy trial. Lancet Oncol. 2005 May;6(5):271-8. doi: 10.1016/S1470-2045(05)70101-7. PMID 15863374
- [Background] Reisinger KS, Block SL, Lazcano E, et al. A randomized controlled trial to evaluate the safety and immunogenicity of a quadrivalent human papillomavirus (types 6, 11, 16, and 18) L1 virus-like particle vaccine in preadolescents and adolescents. The 24th Annual Meeting of the European Society for Paediatric Infectious Diseases; 2006 May 3-5

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited during office visits.
Groups:
- Placebo: Patients who are in the control group will receive a placebo of saline at initial date, 2 months and 6 months.
- Gardasil Group: The treatment group will receive a 0.5 mL intramuscular injection of Gardasil (quadrivalent HPV vaccine) in their upper extremity and again at two months and six months after enrollment.
Period: Overall Study
Arm/Group | Placebo | Gardasil Group
Started | 17 | 15
Completed | 5 | 3
Not Completed | 12 | 12

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were reported (age, gender, region of enrollment). Five of 17 patients in the placebo group completed study follow-up through at least 6 months and received all three study injections. Seven of 15 patients in the Gardasil group completed study follow-up through at least 6 months and received all three study injections.
Groups:
- Placebo: Patients in this group received placebo of saline at initial date, 2 months and 6 months after enrollment.
- Gardasil: Patients in this group received Gardasil injection at initial date, 2 months and 6 months after enrollment.
- Total: Total of all reporting groups
Arm/Group | Placebo | Gardasil | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 15 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (10) | 37 (13) | 37 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  United States | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of This Study is Persistence and Recurrence of Anal Warts as Compared Between the Experimental and Control Groups.
Description: Persistence of anal warts will be measured by the presence of any lesions at one month follow-up after surgery. Recurrence of anal warts will be measured by the development of new lesions after one month of follow-up.
Time Frame: Follow up evaluation after treatment at 1, 3, 6, 9. 12, 15, 18 months after initial treatment
Population: Five patients from the placebo group and seven patients from the gardasil group completed all three injections per the protocol. The remaining patients did not complete study-required follow-up and therefore could not be analyzed. One patient from the Gardasil Group and one patient from the placebo group met the outcome measure of recurrence.
Measure: Number; unit: participants
Groups:
- Placebo Group: Patients who received placebo of saline at initial visit, 2 months and 6 months after enrollment.
- Gardasil Group: Patients who received Gardasil injection at initial visit, 2 months, and 6 months after enrollment.
Arm/Group | Placebo Group | Gardasil Group
Number analyzed (Participants) | 5 | 7
participants | 1 | 1

ADVERSE EVENTS:
Description: Serious and/or other non-serious adverse events were not collected or assessed.
Groups:
- Placebo: Patients who are in the control group received a placebo of saline at initial date, 2 months and 6 months.
- Treatment Group: The treatment group received a 0.5mL intramuscular injection of Gardasil (quadrivalent HPV vaccine) in their upper extremity and again at two months and six months after enrollment.
Arm/Group | Placebo | Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Compliance with follow up was an ongoing issue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No